CLINICAL TRIAL: NCT06938893
Title: Study on Cardiac Output Evaluation Based on Wearable Monitoring Data
Status: Not yet recruiting | Type: Observational
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: HZKY-PJ-2024-57
Record Dates: First submitted 2025-01-17; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Output
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Exercise — Cardiac output (CO) was measured after exercise intervention in patients with normal cardiac function

SUMMARY:
Based on the monitoring data of wearable devices, with cardiac output (CO) as the gold standard, this study intends to develop a non-invasive evaluation model of CO based on wearable data, and optimize the parameters to realize the cardiac capacity detection function in resting and exercise states on the wearable device.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Left ventricular ejection fraction (Left ventricular ejection fraction, LVEF) < 50%(200 subjects)
* Left ventricular ejection fraction (Left ventricular ejection fraction, LVEF) ≥50% (100 subjects)
* Able to use smart phones and operate wearable devices such as wristbands/watches

Exclusion Criteria:

* Patients with pacemaker implantation
* No smartphone
* Currently participating in other clinical trials
* Lactating women
* Pregnant Women
* Unable to run and ride due to personal physical and external reasons (subjects participating in the exercise state cardiac output model study)
* Physical examination results in the past year have clear cardiovascular, metabolic, bone and joint related diseases that have exercise risk, or have diseases and related potential health risks confirmed by the self-examination form of physical status before exercise (participants in the exercise state cardiac output model study)
* No informed consent was obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two hundred HF patients with an left ventricular ejection fraction (LVEF) of less than 50% and 100 normal cardiac function subjects with an LVEF of 50% or greater were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiac output | From enrollment to the end of follow-up at 1 month
  Taking cardiac function indicators such as cardiac output by echocardiography as the gold standard, using wearable device monitoring data（Photoplethysmographic pulse wave）, the resting state cardiac output artificial intelligence machine learning model was established, and the sensitivity, specificity, positive predictive value, negative predictive value, F1 score, diagnostic efficiency Area Under Curve (AUC), and the sensitivity, specificity, positive predictive value, negative predictive value, F1 score, diagnostic efficiency of the model were calculated. AUC), precision and precision-recall curves were used to evaluate the performance of the model.

SECONDARY OUTCOMES:
Heart failure | From enrollment to the end of follow-up at 1 month
  Heart failure symptoms, acute heart failure episodes, rehospitalization rates, and cardiovascular mortality

IPD SHARING:
Plan to Share IPD: Undecided